CLINICAL TRIAL: NCT00621985
Title: Dexamethasone Treatment of Congenital Adrenal Hyperplasia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Joseph Majzoub, Children's Hospital Boston
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 08-01-0025
Record Dates: First submitted 2008-02-11; First posted 2008-02-22 (Estimated); Results first posted 2011-02-23 (Estimated); Last update posted 2011-02-23 (Estimated); Status verified 2011-01

CONDITIONS: Adrenal Hyperplasia, Congenital
MeSH Terms: conditions — Adrenal Hyperplasia, Congenital | interventions — Dexamethasone; Calcium Dobesilate; Hydrocortisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Experimental (Experimental): Experimental therapy with nocturnal dexamethasone.
  Interventions: Drug: dexamethasone; Drug: Hydrocortisone

INTERVENTIONS:
Drug: dexamethasone — Dexamethasone will be given at a dose that equals 1/50 of the total daily hydrocortisone dose of the patient. It will be given in solution form at 10 PM for 3 days.
  Other Names: Decadron
Drug: Hydrocortisone — Subjects were given their baseline hydrocortisone regimen which was three times daily for 4 of the subjects and twice daily for one subject. Doses were given at 8 AM, 2 PM, and 8 PM. The 2 PM time point was skipped for the subject who received hydrocortisone twice daily. Doses ranged from 6.9 to 18.5 milligrams per meter squared per day and were based on each individual's baseline regimen.

SUMMARY:
The purpose of this study is to determine if dexamethasone given at night is a more effective treatment for congenital adrenal hyperplasia in young children than standard three times per day hydrocortisone. Our hypothesis is that nocturnal dexamethasone will lead to more efficient suppression of the hypothalamic-pituitary-adrenal axis. We performed a cross-over trial comparing hormonal control during two 24-hour hospitalizations, one on hydrocortisone and one on nocturnal dexamethasone.

DETAILED DESCRIPTION:
This is a Phase II clinical trial, intended to estimate the effect of instituting Dexamethasone therapy in comparison to prior standard therapy. Each subject provides his own baseline data. There is no control group. Patients with CAH who meet inclusion criteria will be admitted to the clinical research center for two 24 hour hospitalizations. Adrenal hormone profiles will be measured during each hospitalization. The patient will take his or her baseline hydrocortisone regimen during one hospitalization and a new regimen consisting of a single daily nocturnal dose of Dexamethasone during the second hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* Classic salt-wasting 21-hydroxylase deficient congenital adrenal hyperplasia
* Pre-pubertal children with bone ages below 8 years

Exclusion Criteria:

* Age less than 2 years
* Patients with additional medical conditions necessitating glucocorticoid therapy.
* Patients on phenytoin, barbiturates, and rifampin as these medications accelerate the metabolism of glucocorticoids.
* Patients on ketoconazole as this medication increases the bioavailability of glucocorticoids.

Ages: 2 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 5 (Actual)
Dates: Start 2008-04; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Majzoub, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Children's Hospital Boston, Boston, Massachusetts, United States

REFERENCES:
- [Result] Dauber A, Feldman HA, Majzoub JA. Nocturnal Dexamethasone versus Hydrocortisone for the Treatment of Children with Congenital Adrenal Hyperplasia. Int J Pediatr Endocrinol. 2010;2010:347636. doi: 10.1155/2010/347636. Epub 2010 Sep 14. PMID 20871859

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from the Endocrine Clinic at Children's Hospital Boston from April through November 2008.
Pre-assignment Details: This was a cross over study. All subjects were admitted on their baseline hydrocortisone regimen for a 24 hour hospital admission. They then had a second hospital admission within 8 weeks while being administered the dexamethasone therapy.
Groups:
- Experimental: Baseline hydrocortisone was given at a dose determined by the subject's primary endocrinologist and was given either 2 or 3 times per day as per their home regimen. Experimental therapy with nocturnal dexamethasone given at a dose equivalent to 1/50th of the total daily hydrocortisone dose. This dose was given at 10 PM for three nights with the admission to the hospital occurring on the 3rd day prior to the 3rd evening dose.
Period: Hydrocortisone Admission
Arm/Group | Experimental
Started | 5
Completed | 5
Not Completed | 0
Period: Dexamethasone Admission
Arm/Group | Experimental
Started | 5
Completed | 4
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Groups:
- Experimental Group: These subjects were admitted twice, once while on baseline hydrocortisone and once on dexamethasone.
Arm/Group | Experimental Group
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 5
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Percent Difference in the Mean Log Transformed Area Under the Curve of 17-hydroxyprogesterone Between Regimens
Description: Each subject was admitted for 2 24 hour hospitalizations, one on hydrocortisone and one on dexamethasone. Due to the timing of blood draws, the serum hormonal profile was only measured for 23 hours. The primary outcome was the Percent Difference in the Mean log transformed Area under the curve of 17-hydroxyprogesterone between the two regimens.
Time Frame: 23 hours
Population: Only four participants completed both the hydrocortisone and dexamethasone admissions.
Measure: Log Mean (Standard Deviation); unit: Log Mean Area Under the Curve
Groups:
- Dexamethasone Admission: This is the second admission of the protocol during which the subject received dexamethasone.
- Hydrocortisone Admission: This is the first admission of the protocol during which the subject received hydrocortisone.
Arm/Group | Dexamethasone Admission | Hydrocortisone Admission
Number analyzed (Participants) | 4 | 4
Log Mean Area Under the Curve | 3.16 (0.93) | 3.91 (0.66)
Statistical Analysis 1: Comparison: Dexamethasone Admission vs Hydrocortisone Admission; A t-test was performed comparing the mean long transformed area under the curve of 17-hydroxyprogesterone between the dexamethasone and hydrocortisone arms. The percent difference in mean log AUC was calculated as: (Mean log AUC on dexamethasone - Mean log AUC on hydrocortisone)/Mean log AUC on hydrocortisone; Test type: Superiority or Other; p = 0.09, t-test, 2 sided; Percent Difference = -19

ADVERSE EVENTS:
Arm/Group | Dexamethasone Admission | Hydrocortisone Admission
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 1/5 | 0/5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dexamethasone Admission (N=5) | Hydrocortisone Admission (N=5)
IV infiltration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — IV accidentally placed intrarterially and had to be removed. Study was discontinued for this individual. There was no permanent injury or adverse sequelae.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes